CLINICAL TRIAL: NCT05953103
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Phase II Clinical Trial to Evaluate the Efficacy and Safety of Different Doses of Edaravone Dexborneol Concentrated Solution for Injection Combined With Conventional Medical Therapy in the Treatment of Patients With Cerebral Hemorrhage
Brief Title: Evaluate the Efficacy and Safety of Different Doses of Edaravone Dexborneol Concentrated Solution for Injection Combined With Conventional Medical Therapy in the Treatment of Patients With Cerebral Hemorrhage
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Simcere Pharmaceutical Co., Ltd (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SIM0355-201
Record Dates: First submitted 2023-06-24; First posted 2023-07-19 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-01

CONDITIONS: Subjects With Cerebral Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Part A 1 - Subjects with cerebral hemorrhage (Synbixin 37.5 mg; placebo group ) (Experimental)
  Interventions: Drug: Synbixin/Placebo
- Part A 2 - Subjects with cerebral hemorrhage ( Synbixin 62.5 mg; placebo group ) (Experimental)
  Interventions: Drug: Synbixin/Placebo
- Part B - Subjects with cerebral hemorrhage ( Synbixin TBD mg; placebo group ) (Experimental)
  Interventions: Drug: Synbixin/Placebo

INTERVENTIONS:
Drug: Synbixin/Placebo — Synbixin/Placebo

SUMMARY:
The SIM0355-201 trial is a multicenter, randomized, double-blind, placebo-controlled exploratory clinical trial with the main study objective of evaluating the safety and tolerability of different doses of Edaravone Dexborneol concentrate for injection combined with conventional medical therapy in patients with cerebral hemorrhage. The subject had a clinical diagnosis of cerebral hemorrhage, within 6-24 hours from stroke onset to start of study treatment, with the bleeding site in basal ganglia and a hematoma volume ≤ 30 ml at the bleeding site. The trial was divided into two periods (Period A and Period B), with Period A being a dose escalation period divided into two dose levels: the first dose level group (Dose 1 group: Synbixin 37.5 mg; placebo group) and the second dose level group (Dose 2 group: Synbixin 62.5 mg; placebo group).

DETAILED DESCRIPTION:
The SIM0355-201 trial is a multicenter, randomized, double-blind, placebo-controlled exploratory clinical trial with the main study objective of evaluating the safety and tolerability of different doses of Edaravone Dexborneol concentrate for injection combined with conventional medical therapy in patients with cerebral hemorrhage. The subject had a clinical diagnosis of cerebral hemorrhage, within 6-24 hours from stroke onset to start of study treatment, with the bleeding site in basal ganglia and a hematoma volume ≤ 30 ml at the bleeding site. The trial was divided into two periods (Period A and Period B), with Period A being a dose escalation period divided into two dose levels: the first dose level group (Dose 1 group: Synbixin 37.5 mg; placebo group) and the second dose level group (Dose 2 group: Synbixin 62.5 mg; placebo group). Safety was assessed unblinding after the end of study treatment for all subjects in the first dose level group and escalated to the second dose level if the "safe dose" criterion was met, otherwise the trial was terminated; safety was assessed unblinding after the end of study treatment for all subjects in the second dose level group and the 62.5 mg dose level was selected to enter Stage B if the "safe dose" criterion was met, otherwise the 37.5 mg dose level was selected to enter Stage B.

ELIGIBILITY:
Inclusion Criteria:

1. the subject himself or her legal representative has signed the informed consent form;
2. aged ≥ 18 years and ≤ 80 years, male or female;
3. clinical diagnosis of cerebral hemorrhage, in line with the Chinese Medical Association Neurology Score issued by the "Key Points in the Diagnosis of Various Major Cerebrovascular Diseases in China 2019" cerebral hemorrhage diagnostic criteria [1];
4. the bleeding center site is located in the basal ganglia;
5. intracranial hematoma volume ≤ 30 ml;
6. NIHSS score at enrollment total score ≥ 6 points and ≤ 20 points, and the sum of items 5 and 6 ≥ 2 points;
7. coma degree is mild to moderate, Glasgow Coma Scale (GCS) ≥ 9 points;
8. the time from the onset of this stroke to the start of study treatment is 6 to 24 hours (subjects who sign the informed consent form should receive study treatment as soon as possible, some subjects meet the criteria during the screening period, more than 24 hours when starting study treatment, this patient should terminate the study treatment);
9. mRS score of 0 or 1 before onset.

Exclusion Criteria:

1. allergic to edaravone, dextromethorphan or contained excipients;
2. stroke within the past 3 months;
3. other concomitant sites of hematoma volume > 5ml, or the need for external ventricular drainage of patients with intraventricular hemorrhage;
4. patients with obstructive hydrocephalus;
5. drugs, vascular structural damage or coagulation disorders caused by cerebral hemorrhage;
6. vital signs unstable, suspected cerebral hernia, deep coma or anisocoria and other critical manifestations;
7. after this onset has been applied edaravone or dextromethorphan components (such as edaravone injection, Angong Niuhuang pills, Xingnaojing, etc.) of drugs, or has applied a total of more than 2 times the daily recommended dose of the instructions of the following drugs: citicoline, oxiracetam, piracetam, ulinastatin;
8. planned surgical evacuation of hematoma, including: craniotomy hematoma evacuation, minimally invasive surgery and decompressive craniectomy;
9. ALT or AST > 2.0 × ULN or previously known liver disease, such as acute hepatitis, chronic active hepatitis, cirrhosis, etc., previously known kidney disease, renal insufficiency, serum creatinine > 1.5 × ULN or creatinine clearance < 50 mL/min;
10. Suffering from other bleeding disorders, such as thrombocytopenic purpura, bleeding tendency caused by vascular injury, hemophilia and other coagulation disorders, gastrointestinal ulcers, urinary tract bleeding, hemoptysis, etc.;
11. Presence of severe, progressive, or uncontrolled symptoms of renal, hepatic, hematological, gastrointestinal, pulmonary, cardiovascular, neurological, or cerebral disease that, in the opinion of the investigator, place the subject at unacceptable risk by participating in this study;
12. With severe active bacterial or viral infection;
13. Concurrent malignancy or ongoing anti-tumor therapy;
14. With severe systemic disease, expected survival < 90 days;
15. Patients with severe mental disorders and dementia;
16. Patients who are pregnant, lactating and planning pregnancy;
17. Reasons for other investigators' unsuitability to participate in this trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380 (Estimated)
Dates: Start 2023-07-03 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of serious adverse events (SAEs) up to 90 days after the first dose of treatment | up to 90 days after the first dose of treatment

SECONDARY OUTCOMES:
Incidence of deaths up to 90 days after the first dose of treatment | up to 90 days after the first dose of treatment
Proportion of subjects with AEs, AEs leading to dose interruption or discontinuation, AEs related to study drug, AEs of special interest (AESls), and with abnormal vital signs, abnormal physical examination findings and abnormal laboratory tests results | up to 90 days after the first dose of treatment
Proportion of subjects with modified Rankin Score (mRS) 0-2, which assesses the degree of disability or dependence in daily activities, with scores ranging from 0 (no symptoms) to 6 (death), at 90 days after the first dose of treatment | at 90 days after the first dose of treatment
Proportion of subjects with modified Rankin Score (mRS) 0-1, which assesses the degree of disability or dependence in daily activities, with scores ranging from 0 (no symptoms) to 6 (death), at 90 days after the first dose of treatment | at 90 days after the first dose of treatment
Distribution of subjects with modified Rankin Score (mRS), which assesses the degree of disability or dependence in daily activities, with scores ranging from 0 (no symptoms) to 6 (death), at 14, 30, 90 days after the first dose of treatment | at 14, 30, 90 days after the first dose of treatment
Distribution of subjects with Glasgow Outcome Score (GOS), which measures functional outcome, with scores ranging from I (Dead) to V (Good Recovery), at 14, 30, 90 days after the first dose of treatment | at 14, 30, 90 days after the first dose of treatment
Change from baseline in National Institutes of Health Stroke Scale (NIHSS), which quantifies the impairment caused by a stroke, with scores ranging from 0 (no stroke symptoms) to 42 (the most severe stroke) | at 14, 30, 90 days after the first dose of treatment
Proportion of subjects with National Institutes of Health Stroke Scale (NIHSS) 0-2, which quantifies the impairment caused by a stroke, with scores ranging from 0 (no stroke symptoms) to 42 (the most severe stroke) | at 14, 30, 90 days after the first dose of treatment
Proportion of subjects with Barthel index (BI), which measures a person's ability to complete activities of daily, with scores ranging from 0 (fully dependent) to 20 (fully independent), at 90 days after the first dose of treatment | at 90 days after the first dose of treatment
Imaging endpoints：Change from baseline in perihematomal edema volume (PHEv) and hematoma volume (HV) in milliliters | at 3, 7, 14 days after the first dose of treatment
Imaging endpoints：Change from baseline in edema extension distance (EED) in millimetres c) Change from baseline in relative perihematomal edema (PHEv/Hv) in odds ratio | at 3, 7, 14 days after the first dose of treatment
Imaging endpoints: Change from baseline in relative perihematomal edema (PHEv/Hv) in odds ratio | at 3, 7, 14 days after the first dose of treatment
Plasma pharmacokinetic endpoints: Cmax: maximum observed plasma concentration for edaravone and dexborneol | 1 hour pre-dose and 1, 2 hour post-dose at 3, 14 days after the first dose of treatment
Plasma pharmacokinetic endpoints: Tmax: time to reach the maximum plasma concentration (Cmax) for edaravone and dexborneol | 1 hour pre-dose and 1, 2 hour post-dose at 3, 14 days after the first dose of treatment
Plasma pharmacokinetic endpoints: AUC(0-inf): area under the plasma concentration-time curve from time 0 to infinity for edaravone and dexborneol | 1 hour pre-dose and 1, 2 hour post-dose at 3, 14 days after the first dose of treatment
Plasma biomarker endpoints: a) Change from baseline in white blood cell count (WBC) in 109/L; b) Change from baseline in C-reactive protein (CRP), Thioredoxin (TRX) and matrix metalloproteinases (MMP) in mg/L | at 3, 7, 14 days after the first dose of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Xiaonan Yao, Study Director — Simcere Pharmaceutical Co., Ltd
Locations (1):
- The First Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No